CLINICAL TRIAL: NCT07312019
Title: Optimization of Medical Time in the Emergency Department: Impact of an AI-Based System on Prescription Entry
Acronym: YGénHIAL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Centre Hospitalier Public du Cotentin (Unknown); University Hospital, Bordeaux (Other); University Hospital, Strasbourg, France (Other); Clinique de l'Estrée (Unknown); CHU Aix-en-Provence (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PI2024_843_0120
Record Dates: First submitted 2025-11-17; First posted 2025-12-31 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Drug-related Iatrogenesis; Emergency Department; Artificial Intelligence; Clinical Decision Support; Prescription; Transcription; Medication; Reconciliation
Keywords: Drug-related iatrogenesis; emergency department; artificial intelligence; clinical decision support; randomized trial; medication; reconciliation; prescription; transcription
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard prescription (Active Comparator): Standard prescription management
  Interventions: Other: current hospital-standard databases
- PoSOS (Experimental): POSOS-assisted prescription management
  Interventions: Device: Posos

INTERVENTIONS:
Other: current hospital-standard databases — Prescription management using current hospital-standard databases and tools
  Arms: Standard prescription
Device: Posos — Prescription management supported by POSOS device (OCR+AI) for structured data entry and clinical decision support
  Arms: PoSOS

SUMMARY:
Drug-related iatrogenesis is a major public health issue, accounting for a significant proportion of adverse events and hospitalizations in emergency departments. Optimizing prescription management in this context is critical to improve both patient safety and physician efficiency This study aims to evaluate the impact of the POSOS AI-driven device on the medical time required for prescription management in polymedicated patients admitted to emergency departments. The main objective is to establish whether the use of POSOS can reduce transcription time compared to standard electronic management.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Admission to emergency department at a participating center
* Polymedicated patients with prescriptions including ≥8 medication lines (including those for long-term illnesses)
* Signed informed consent

Exclusion Criteria:

* Patient under legal protection/judicial measures (guardianship/custody)
* Lack of signed informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 770 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Medical time required for the transcription of prescriptions | Day 1
  Medical time required for the transcription of prescriptions for at-risk polymedicated patients at emergency admission. This is measured by the duration needed to transcribe prescriptions into the structured electronic health record by physicians, assessed by direct observation with a stopwatch

SECONDARY OUTCOMES:
Number of drug-related problems (DRPs) identified per patient | day 1
Proportion and type of transcription errors (medication name or dosage) | day 1
Identification of DRPs by subtype and severity | day 1
Rate of reconciled medication histories and structured documentation | day 1
Time delays between triage, anamnesis, and diagnosis | day 1
Length of emergency department stay and downstream hospitalizations | day 1
Readmission rates | at 3 months
Overall survival | at 6 months
Mapping of DRPs by subtype and severity | day 1

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No